CLINICAL TRIAL: NCT00582868
Title: Brain Oxygen Tension Level, Cerebral Perfusion and Cleaved-tau Protein for Detection of Cerebral Vasospasm and Independent Predictor of Poor Outcome After Aneurysmal Subarachnoid Hemorrhage
Brief Title: Use of Brain Oxygen Tension Level and Cleaved-tau Protein to Detect Vasospasm After SAH
Status: Terminated | Type: Observational
Why Stopped: Insufficient subject enrollment
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: H-2006-0421
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2012-04

CONDITIONS: Subarachnoid Hemorrhage; Cerebral Vasospasm
Keywords: Subarachnoid hemorrhage; Cerebral Vasospasm; Cleaved-tau protein; Brain oxygen tension level
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cerebrospinal fluid Whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hemorrhage: Patients having experienced subarachnoid hemorrhage and have in place a ventriculostomy
  Interventions: Device: Licox Brain Oxygen Monitor; Other: CSF; Other: Whole blood

INTERVENTIONS:
Device: Licox Brain Oxygen Monitor — use of data from brain oxygen monitor for analysis
Other: CSF — analysis of CSF for cleaved tau protein
Other: Whole blood — Analysis of whole blood for cleaved-tau protein

SUMMARY:
The purpose of this study is to investigate if brain oxygen levels, levels of a specific protein in the cerebrospinal fluid and blood (Cleaved-tau protein), and brain blood flow can predict spasm of brain blood vessels after bleeding in the brain from a ruptured aneurysm.

DETAILED DESCRIPTION:
Rupture of a cerebral aneurysm causes subarachnoid hemorrhage (SAH). Blood in the subarachnoid space of the brain can cause irritation of the cerebral blood vessels, leading to constriction of these vessels, a phenomenon known.as vasospasm. Cerebral vasospasm can cause stroke and possibly death. Of all the patients with SAH, approximately 20-40% will suffer from clinical vasospasm and more than 60% of those patients will never get back to their previous functional status. Tools to identify early vasospasm and thus early treatment could greatly decrease the morbidity and mortality following SAH.

Cleaved tau protein is a neuronal marker that has been detected in blood and CSF of stroke patients early in its time course. Since vasospasm can lead to stroke, the purpose of this project is to determine whether increase in cleaved tau protein in blood and/or CSF can predict early stroke from vasospasm. Changes in brain oxygen tension measured by a brain tissue oxygen monitor and cerebral blood flow measured by CT perfusion will be correlated with cleaved tau protein levels and clinical status. Utilizing statistical analysis the levels of Cleaved tau protein, brain oxygen and blood flow during hospitalization will be correlated with patient outcome. Through this study we hope to identify increase in cleaved tau protein and decrease in cerebral blood flow and oxygenation as predictors of early vasospasm. Early detection and treatment of vasospasm could decrease the stroke rate in SAH patients and therefore be of great benefit to society.

ELIGIBILITY:
Inclusion Criteria:

* Patients with subarachnoid hemorrhage
* Patients with external ventricular drains

Exclusion Criteria:

* Patients in whom consent is not attainable

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with subarachnoid hemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2007-05; Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Changes in brain oxygen tension level, cerebral blood flow, and cleaved tau protein levels in correlation to cerebral vasospasm | The first 14 days after subarachnoid hemorrhage

SECONDARY OUTCOMES:
Clinical outcome score correlated to changes in brain oxygen tension level, cerebral blood flow, and cleaved tau protein levels | Three months after subarachnoid hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Baskaya, MD, Principal Investigator — University of Wisconsin Department of Neurosurgery; Bobby M Agrawal, MD, Principal Investigator — University of Wisconsin Department of Neurosurgery
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States